CLINICAL TRIAL: NCT01127126
Title: Treatment of the Overactive Bladder in Postmenopausal Women With Bryophyllum Pinnatum Versus Placebo (a Multicenter, Prospective, Double-blind Randomised, Placebo-controlled Clinical Pilot Study, Phase II Drug Study)
Brief Title: Bryophyllum Versus Placebo for Overactive Bladder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2009-0075/4
Record Dates: First submitted 2010-05-17; First posted 2010-05-20 (Estimated); Last update posted 2012-01-19 (Estimated); Status verified 2012-01

CONDITIONS: Overactive Bladder
MeSH Terms: conditions — Urinary Bladder, Overactive

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Bryophyllum (Active Comparator): muscle relaxing substance
  Interventions: Drug: Bryophyllum pinnatum, Placebo in form of Lactose
- Placebo (Placebo Comparator): control group postmenopausal women suffering from overactive bladder
  Interventions: Drug: Bryophyllum pinnatum, Placebo in form of Lactose

INTERVENTIONS:
Drug: Bryophyllum pinnatum, Placebo in form of Lactose — Comparison Bryophyllum (2100mg/d) against Placebo (2100mg/d) regarding effectivity and safety.
  Bryophyllum and Placebo are both administered for 8 weeks. Bryophyllum and Placebo are both given in form of capsules, 350mg per capsule, 2-2-2/d.
  Other Names: Bryophyllum pinnatum/Kalanchoe; Lactose/milk sugar

SUMMARY:
E: The pharmacological effect of Bryophyllum pinnatum could be shown on uterine smooth muscle cells, on spontaneous and oxytocin-stimulated contractions. Smooth muscle relaxation is not only required for preventing premature labour but also for symptom's relief of overactive bladder (OAB). According to previous preclinical and clinical studies, an inhibiting effect of Bryophyllum on OAB is assumed.

20 women are included in this phase 2 drug study, treated with Bryophyllum pinnatum in form of the commercially available Bryophyllum tablets into capsules (verum: 3x2capsules/day) or lactose capsules (placebo: 3x2 capsules/day), 10 women in each group. Duration of the drug administration is 8 weeks.

Primary endpoint is the reduction of micturitions per 24 hours (measured by filling in a voiding dairy), secondary endpoints are the improvement of quality of life (measured by using the King's Health Questionnaire and the ICIQ-OAB, two questionnaires, validated for the german language, for women with incontinence), increase of the micturition volumes and reduction of urge episodes (measured by the patients and recorded in a voiding dairy) and the registration of adverse events during the study phase. Ethics committee approval has been given 10th March 2010. - Trial with medicinal product

DETAILED DESCRIPTION:
In the therapeutic concept of the treatment of OAB, antimuscarinic drugs play a central role. Antimuscarinics are known to inhibit the contraction of detrusor muscle (smooth muscle cells) and block the muscarinic receptor (M2/M3) important for efferent nerve conduction. This conventional therapy for OAB can have important adverse effects, notably on the gastrointestinal tract with constipation, on the excretory glands in the sense of xerostomia/xerophthalmia, on the nerve cells of the brain inhibiting cognitive function and in the heart muscle cells accelerating the heart rate. Especially elderly people are affected by these undesirable effects. Because of changes in the receptor profile, the effect of antimuscarinics and improvement of symptoms might be lowered in elderly people and another substance with less side effects would be of great interest. No such adverse effects are reported for B. pinnatum. Until now, there are no data for its use in OAB. Efficacy and tolerability of B. pinnatum in the treatment of OAB are the major outcome measures of this clinical trial.

* 20 women are included in this phase 2 drug study, treated with Bryophyllum pinnatum in form of the commercially available Bryophyllum tablets into capsules (verum: 3x2capsules/day) or lactose capsules (placebo: 3x2 capsules/day), 10 women in each group. Recruitment time is planned from July 2010 to June 2011.
* Duration of the drug administration is 8 weeks.
* Primary endpoint is the reduction of micturitions per 24 hours (measured by filling in a voiding dairy)
* secondary endpoints are the improvement of quality of life (measured by using the King's Health Questionnaire and the ICIQ-OAB, two questionnaires, validated for the german language, for women with incontinence), increase of the micturition volumes and reduction of urge episodes (measured by the patients and recorded in a voiding dairy) and the registration of adverse events during the study phase. Ethics committee decision has been given.

ELIGIBILITY:
Inclusion criteria:

* postmenopausal women with OAB
* prior cystoscopy to exclude a malignancy
* local or systemic hormone restitution therapy is allowed
* prior incontinence operation (if the operation dates back more than 12 months)
* german or french speaking patients and a given informed consent

Exclusion criteria:

* Intolerance against a substance or a compound
* participation in an other study 4 weeks prior to inclusion
* urinary tract infection
* drug abuse
* bladder affecting drugs like anticholinergics, diuretics, muscle relaxing medicaments and phytotherapeutics
* lactose intolerance
* diabetes mellitus.

Ages: 18 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2010-12; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Reduction of micturition frequency/24h | micturition protocol three days before baseline visit and follow-up control 2 and 8 weeks after medication intake and 6 weeks after the completed medication period
  micturition frequency measured with the micturition protocoll

SECONDARY OUTCOMES:
quality of life | before baseline control, at follow-up control 8 weeks after begin of medication intake and 6 weeks after end of medication intake
  quality of life is measured by the King's Health Questionnaire and the ICIQ-OAB, a specific questionnaire for OAB
safety of Bryophyllum intake and adverse events | during medication intake at 2 weeks and 8 weeks after start of medicaton intake, measured by a personal adverse event protocol
  Number of Participants with Adverse Events as a Measure of Safety and Tolerability

CONTACTS AND LOCATIONS:
Overall Officials: 01 Studienregister MasterAdmins, Study Director — UniversitaetsSpital Zuerich
Locations (1):
- Department of Obstetrics and Gynecology, Zurich, Switzerland

REFERENCES:
- [Derived] Betschart C, von Mandach U, Seifert B, Scheiner D, Perucchini D, Fink D, Geissbuhler V. Randomized, double-blind placebo-controlled trial with Bryophyllum pinnatum versus placebo for the treatment of overactive bladder in postmenopausal women. Phytomedicine. 2013 Feb 15;20(3-4):351-8. doi: 10.1016/j.phymed.2012.10.007. Epub 2012 Dec 4. PMID 23218404